CLINICAL TRIAL: NCT07212673
Title: Combining Digital Cognitive-behavior Therapy With Mindfulness Training for Binge Eating Disorder: a Feasibility Randomized Controlled Trial
Brief Title: Combining Digital Cognitive-behavior Therapy With Mindfulness Training for Binge Eating Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yeshiva University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Margaret Sala, Assistant Professor, Yeshiva University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20251574; K23AT012126 (NIH)
Record Dates: First submitted 2025-09-17; First posted 2025-10-08 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Binge Eating Disorder
Keywords: binge eating; eating disorder; obesity
MeSH Terms: conditions — Binge-Eating Disorder; Bulimia; Feeding and Eating Disorders; Obesity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT-based Mindful Courage + Coached Self-Monitoring (Experimental): CBT-based Mindful Courage is a digital intervention including mindfulness and CBT elements for individuals with binge eating disorder. It will consist of 16 self-guided modules. Elements included in the intervention include psychoeducation, self-monitoring, regular eating, goal-setting, weekly weighing, eating a sufficient amount of food at each meal, eating a range of foods reduction of overvaluation of weight and shape, addressing shape/body checking or avoidance, behavior chain analysis, problem solving, awareness and acceptance of binge eating urges, thoughts and emotions, values awareness, values clarification, values-based decision making, self-compassion, exploring needs underlying binge eating urges, mindful eating, hunger and fullness awareness, self-compassion, and self-care. Weekly mindfulness practice (at least 3x per week) is heavily emphasized. Participants will also be asked to self-monitor their food intake in Recovery Record and will receive phone coaching.
  Interventions: Behavioral: CBT-based Mindful Courage; Behavioral: Coached Self-Monitoring
- Coached Self-Monitoring (Active Comparator): Participants will be asked to self-monitor their food intake in Recovery Record and will receive phone coaching
  Interventions: Behavioral: Coached Self-Monitoring

INTERVENTIONS:
Behavioral: CBT-based Mindful Courage — Self-guided online intervention
  Arms: CBT-based Mindful Courage + Coached Self-Monitoring
Behavioral: Coached Self-Monitoring — Participants will log meals in recovery record

SUMMARY:
The investigators will evaluate the acceptability and feasibility of a 16-session digital mindfulness-based and cognitive behavioral therapy (CBT) intervention for binge eating disorder (BED) + coached self-monitoring vs. a coached self-monitoring intervention. This study is a pilot randomized controlled trial.

DETAILED DESCRIPTION:
Procedures include completing: (1) pre-intervention screening assessment; (2) an initial baseline visit; (3) the assigned intervention; (4) a mid-study visit; (5) a post-intervention assessment (~18-weeks after baseline); and (6) a 2-month follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* ability to speak English fluently
* meeting DSM-5 criteria for current BED (i.e., in the past three months)
* willing and able to commit to the entire study protocol

Exclusion Criteria:

* a BMI below 18.5
* requiring immediate treatment for medical complications
* having current anorexia or bulimia nervosa or purging behaviors within the past year
* being pregnant or breast-feeding
* experiencing other severe psychopathology or medical illness that would limit the participants' ability to comply with the demands of the current study (e.g. active suicidal risk, active psychotic disorder, unmedicated bipolar disorder, severe substance use disorder, cancer)
* currently receiving BED or weight loss treatment (treatment for other conditions will be allowed, as long as the treatment is not mindfulness-based)
* currently taking medications for weight loss, or beginning medications that affect eating/weight within the last six months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-02 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility / Completion (questionnaire developed by our lab) | From baseline to 2-month follow-up visit
  Number of participants completing intervention
Acceptability | After completing intervention, an average of 18-weeks
  Dimensions of usability from the System Usability Scale; single-items measuring dimensions of acceptability, including overall satisfaction, engagement, visual appeal of content, understandability of program content, desire to continue the program, perceived skill acquisition, perceived confidence in implementing skills, and perceived helpfulness. Scores for each item range from 1 to 5, with higher scores indicating better acceptability. Scores will be averaged to obtain acceptability ratings.

CONTACTS AND LOCATIONS:
Locations (1):
- Yeshiva University, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No